CLINICAL TRIAL: NCT04538508
Title: Short Term Efficacy of the Combination of Radiofrecuency Diathermy and Supervised Exercise Versus Supervised Exercise Alone in the Treatment of Patellofemoral Pain Syndrome.
Brief Title: Radiofrecuency and Supervised Exercise Versus Supervised Exercise in the Treatment of Patellofemoral Pain Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: University of Seville (Other); Andaluz Health Service (Other Government); Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Alfonso Javier Ibáñez-Vera, Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFPS US
Record Dates: First submitted 2020-08-25; First posted 2020-09-04 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; knee pain; diathermy
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Fever | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not be aware about the treatment any participants will/had received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diathermy (Experimental): Participants that receive 10 sessions of radiofrequency diathermy of 12 minutes of duration
  Interventions: Device: Diathermy; Other: Supervised knee exercises
- Control (Active Comparator): Participants that perform supervised exercises for three weeks
  Interventions: Other: Supervised knee exercises

INTERVENTIONS:
Device: Diathermy — 10 sessions of 12 minutes of radiofrequency diathermy at the anterior surface of the knee, in constant movement
  Arms: Diathermy
Other: Supervised knee exercises — Daily hamstrings exercises, quadriceps exercises and hip exercises, 20 minutes of duration.

SUMMARY:
This study will analyze the effects of a non-invasive radiofrequency diathermy device added to knee exercises on the symptoms of patellofemoral pain syndrome. For this aim, a randomized clinical trial will be carried out with a control group that will perform supervised exercises and an experimental group that will add radiofrequency diathermy to supervised exercises. Diathermy treatment will be performed along three weeks, ten treatment sessions in total, while supervised exercises will be performed daily.

Outcomes to measure will include pain, knee function and quality of life

DETAILED DESCRIPTION:
At first, a meeting will be held with the patients under study where they will be informed and any doubts that may arise in relation to the investigation will be resolved. In addition, the correct adaptation of these to the inclusion and exclusion criteria of our study will be verified. Subsequently, they will be given individually the informed consent prepared expressly for the present study, the doubts arising with respect to this one will be resolved and their signature will proceed. At this time, and individually again, we will proceed to the development of the Clinical History of Physiotherapy where only the information necessary for our study will be collected. To emphasize in this point that the participants will grant their consent for the treatment of the data obtained for scientific purposes, according to the legal norms.

Next, the patients will be randomly assigned to two groups: control group and experimental group. The randomization of the sample was done through the EPIDAT software in version 3.1 between the Experimental Group and the Control Group. Subsequently, the evaluations and measurements of the study variables will be carried out by the research team.

CONTROL GROUP: them will be provided exclusively therapeutic exercises protocol that you must be performed supervised by a physiotherapist following a daily activity for three weeks.

EXPERIMENTAL GROUP: After the initial evaluation, the first 10 treatment sessions will be developed at the rate of five daily sessions in the first week, three sessions on alternate days in the second week and two sessions on alternate days in the third week (3 weeks in total), applying the monopolar dielectric diathermy by radiofrequency in the anterior aspect of the knee, in dynamic application in one of the members: affect or randomized (uni or bilateral pathology, respectively). This diathermy will be combined with the same supervised therapeutic exercise program of the control group.

The treatment is administered with a pulsed non-invasive radiofrequency device with 30V peak power along 12 minutes, with a dose submitis (grade I) for three weeks. The first week, daily treatment will be perform from Monday to Friday, second week on Monday, Wednesday and Friday and the third week on Monday and Thursday.

After the tenth treatment session, all the measurements will be repeated following the same environmental conditions as at the beginning and by the evaluators themselves to the components of both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with patellofemoral pain syndrome more than 6 months old.
* Have an age between 18 years and 50 years.
* Adult patients with anterior knee pain were referred by a primary care physician at a public health center in southern Spain. Those participants with a self-reported pain intensity = 30 mm on the Visual Analog Scale (VAS) and a score <45 points in personal psychology The Apprehension Scale (PPAS) [bathrobe 2017], were invited to participate. The PPAS is a valid, reliable and easy-to-use tool for assessing the apprehension of subjects to receive electrical stimulation therapy [bathrobe 2005].

Exclusion Criteria:

* Any contraindication for the use of MDR
* Present cognitive alterations.
* Have undergone conservative or surgical treatment of the knee in less than 6 months.
* Having received injections of corticosteroids or hyaluronic acid; impaired cognition or communication; and be involved in an ongoing medical-legal dispute.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Knee pain | Baseline
  The perception of pain through the Visual Analogue Scale (EVA). This variable has been obtained through a validated scale of 10 centimeters (0-10), where the subject self-positioned from absence of pain to the worst bearable pain
Knee pain | Three weeks after there first session of treatment
  The perception of pain through the Visual Analogue Scale (EVA). This variable has been obtained through a validated scale of 10 centimeters (0-10), where the subject self-positioned from absence of pain to the worst bearable pain

SECONDARY OUTCOMES:
Knee functional disability | Baseline
  The functional disability, quantified by means of the tests: Kujala Score. This score goes from 0 (high disability) to 100 (no disability)
Knee functional disability | Three weeks after there first session of treatment
  The functional disability, quantified by means of the tests: Kujala Score. This score goes from 0 (high disability) to 100 (no disability)
Knee function | Baseline
  Functional Scale of the Lower Extremity (LEFS). The score goes from 0 (low function) to 80 (great function)
Knee function | Three weeks after there first session of treatment
  Functional Scale of the Lower Extremity (LEFS). The score goes from 0 (low function) to 80 (great function)
Knee flexion range of movement | Baseline
  Active knee joint range of movement. Knee range of movements goes from -10º to 150º
Knee flexion range of movement | Three weeks after there first session of treatment
  Active knee joint range of movement. Knee range of movements goes from -10º to 150º
Knee extension range of movement | Baseline
  Active knee joint range of movement. Knee range of movements goes from -10º to 150º
Knee extension range of movement | Three weeks after there first session of treatment
  Active knee joint range of movement. Knee range of movements goes from -10º to 150º

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Albornoz-Cabello, PhD, Principal Investigator — University of Seville
Locations (1):
- Centro de Salud San José de la Rinconada, San José de la Rinconada, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
Participants did not allow to share their data